CLINICAL TRIAL: NCT07244952
Title: Effects of Vojta Therapy on Posture and Trunk Control in Patients With Sub-acute Stroke
Brief Title: Effects of Vojta Therapy on Posture and Trunk Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Wajeeha Mahmood, Dr, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOL/IREB/25/12/0031
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Stroke; Stroke Ischemic
Keywords: Stroke; cerebral vascular accident; Vojta therapy; pose estimation; posture control; trunk control; upper extremity function
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Vojta therapy and routine physical therapy
  Interventions: Other: Vojta therapy; Other: Routine physical therapy
- Conventional therapy arm (Active Comparator): Routine physical therapy
  Interventions: Other: Routine physical therapy

INTERVENTIONS:
Other: Vojta therapy — Vojta therapy will be implemented for reflex rolling and reflex creeping. A small pressure with dorsal, medial and cranial directional stimuli will be provided. After stimulation the reactions are extension of spine, flexion of hip joint, then knee joint and in the end at ankle joint. 5 sessions per week with a 60-minute session are part of protocol for routine physical therapy and vojta therapy for 8 weeks.
  Other Names: Reflex locomotion therapy
  Arms: Experimental arm
Other: Routine physical therapy — The control group will receive routine physical therapy treatment which will consist of positioning, passive movements of the limbs, sensorimotor exercises for the affected limb using task-oriented training and motor relearning program consisting of repetitive motor skills consisting of functional tasks and involves task breakdown, such as transfers, upper limb function will be performed. 5 sessions per week with a 60-minute session are part of protocol for routine physical therapy and core stability for 8 weeks.

SUMMARY:
Vojta therapy that is reflex locomotion therapy is a neurophysiological rehabilitation approach that stimulates specific "reflex zones" on the body to activate global, innate movement patterns. In stroke rehabilitation, it is used to improve postural control, trunk stability, and functional movement by engaging automatic motor responses. Vojta stimulation can activate motor cortical and subcortical areas as well as postural muscles. Pose estimation will be used to analyze human motion in stroke patients. The study will identify if there is significant difference in the comparative effects of Vojta therapy in addition to routine physical therapy on posture, trunk control and upper extremity motor function in sub-acute stroke patients

DETAILED DESCRIPTION:
Vojta therapy can be used in the early stages of stroke patients' rehabilitation because acute stroke patients are characterized by a disruption in their capacity to react to changes in body posture, necessitating automatic postural adjustment. This study will determine the comparative effects of Vojta therapy in addition to routine physical therapy on posture, trunk control and upper extremity motor function in patients with sub-acute stroke. Body angles will be measured used Vojta therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-65 years
* Both males and females
* First time subacute stroke (7 days post stroke to 3 months)
* Brunnstrom stage 1,2
* A confirmed CT scan for subacute ischemic stroke
* A hemiplegia with score of ≤2 of medical research council scale for muscle strength of the arm (MRCS)
* Premorbid modified Rankin scale score ≤ 3
* Stroke patient who can achieve supported standing
* Patients having NIHSS score 16-20 will be included
* Patient who can achieve sitting for 30 seconds

Exclusion Criteria:

* Severe cognitive impairments that can hinder rehabilitation
* Limitations in communication due to aphasia
* Altered consciousness or dementia (Epple et al., 2020b)
* Patients suffering from postural hypotension

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Posture control | 8 weeks
  To measure posture control posture assessment scale for stroke will be used. It will determine posture after stroke in sitting, standing and lying position. It's a 4-point scale and ranges from 0-36. It consists of 12 items where items are scored from 0-3.It will measure balance in sitting, standing and lying. It will measure the ability of the individual to maintain balance with different positions. Inter ratter reliability for individual items is α=0.88. It has excellent predictive validity with α=0.86
Trunk control | 8 weeks
  Trunk performance will be assessed with Trunk control test. It consists of four items assessed on a three-point ordinal scale. Items include rolling to affected and non-affected side, sitting, and balance in the sitting position for 30 seconds. The total score is from 0 to 100, a higher score of 50 points indicates better performance. A 12-point score indicates abnormal pattern of movement while a 25 -point score means movement was normal. Internal validity is a= o.86 while r= 0.76 It is a validated test for posture control and motor
Motor Evaluation Scale for upper extremity | 8 weeks
  Motor evaluation scale for upper extremity will be used to measure motor activity of arm and hand. It has 8 tasks for arm with six categories of responses and hand has 6 tasks items with three categories. While functional tasks have three items with three categories. It has items of arm with total score of 40 and hand items with total score of 18. The maximum score for the scale is 58. The scale has good test-retest reliability. Reliability is 0.99 for MESUPES arm and 0.97 for MESUPES hand. Validity is 0.87
Pose estimation | 8 weeks
  Pose estimation software will be used for posture information. It will use key points as joints from the body and their position in space and time. In pose estimation the position of each body joint is estimated. It is based on activity recognition. The recognition is done by segmenting the position of the key points of the joints of the individuals in the scene. The Smart phone cameras are used for picture and then the software recognizes the key points on the picture. The software will record precise posture information. The program uses user-selected images to determine angles between various body components

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Wajeeha Mahmood (PT), Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No